CLINICAL TRIAL: NCT02773329
Title: Managing Chemotherapy Induced Neuropathy in Cancer Patients Using Game-based Exercise
Brief Title: Using Game-based Exercise to Improve Balance in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-38347
Record Dates: First submitted 2016-05-09; First posted 2016-05-16 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy; Cancer
Keywords: chemotherapy induced peripheral neuropathy; Cancer; game-based exercise; exercise; wearable sensors; balance; falls; virtual reality
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exergaming; Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention with game-based exercise (Experimental): Subjects will be receiving sensor-based interactive exercise program (game-based exercise) intervention twice a week for 6 weeks.
  Interventions: Other: sensor-based interactive exercise (game-based exercise)
- Intervention without game-based exercise (Active Comparator): Subjects will be receiving non-technology based foot and ankle exercise twice a week for 6 weeks
  Interventions: Other: Intervention without game-based exercise

INTERVENTIONS:
Other: sensor-based interactive exercise (game-based exercise) — This intervention includes interactive game-based balance training including repetitive weight shifting and virtual obstacle crossing tasks. Wearable sensors will provide real-time visual/auditory feedback from foot and ankle position and allowed perception of motor-errors during each motor-action.
  Other Names: virtual reality exercise
  Arms: Intervention with game-based exercise
Other: Intervention without game-based exercise — Subjects are asked to perform non-technology based foot and ankle exercises, which include body weight shifting and obstacle crossing tasks.
  Other Names: non-technology based exercise
  Arms: Intervention without game-based exercise

SUMMARY:
Cancer patients with chemotherapy-induced peripheral neuropathy (CIPN) have deficits in sensory and motor skills leading to inappropriate proprioceptive feedback, impaired postural control and high fall risk. This study will investigate the acceptability and effect of an interactive motor adaptation balance training program based on wearable sensors for improving balance in older cancer patients with CIPN. Cancer patients with confirmed CIPN will be recruited and will be randomized to either intervention (IG) or control (CG) group and followed for 6 months. The intervention group will take part in a 6-week balance training program twice per week in either their home or in clinic (based on subject preference) under the supervision of a qualified research staff member. This intervention includes interactive game-based balance training including repetitive weight shifting and virtual obstacle crossing tasks. Wearable sensors will provide real-time visual/auditory feedback from foot and ankle position and allowed perception of motor-errors during each motor-action. The control group will be instructed to complete a supervised foot and ankle exercise without using sensor technology. Changes in balance, gait, and physical activity, and number of falls will be compared pre- and post-intervention, as well as 3 and 6 month post intervention. Investigators hypothesize that patients receiving sensor-based exercise training will benefit more compared to group receiving conventional non-technology home-based training in terms of improving functional performance and reducing falls.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients
* Men or women aged 55 years or older
* Patients undergoing neurotoxic chemotherapy (agents including platinums, vinca alkaloids, taxanes, proteasome inhibitors and interferons)
* Confirmed peripheral neuropathy (VPT>25) will be eligible to participate

Exclusion Criteria:

* Subjects will be excluded if they have undergone surgery in the last 6-8 weeks
* Have Parkinson's Disease
* Stroke patients
* Dementia patients
* Have an active foot ulcer
* Have an active infection
* Lower extremity major amputation
* Patient is taking medications unrelated to cancer treatment that may affect balance and gait
* Patient has other medical conditions that may affect their balance and gait
* Patient is unable to ambulate without assistance.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Gait Speed change from Baseline to 6 weeks, three months and six months | Baseline, 6 weeks, three months, six months
  walking ability is quantified by gait speed.
Balance change from Baseline to 6 weeks, three months and six months | Baseline, 6 weeks, three months, six months
  balance is quantified by body sway

SECONDARY OUTCOMES:
Fear of falling change from Baseline to 6 weeks | Baseline and 6 weeks
  Measuring fear of falling using Fall Efficacy Scale International (FES-I) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only de-identified data and associated results will be published in peer-review papers or scientific abstracts.

REFERENCES:
- [Result] Schwenk M, Grewal GS, Holloway D, Muchna A, Garland L, Najafi B. Interactive Sensor-Based Balance Training in Older Cancer Patients with Chemotherapy-Induced Peripheral Neuropathy: A Randomized Controlled Trial. Gerontology. 2016;62(5):553-63. doi: 10.1159/000442253. Epub 2015 Dec 18. PMID 26678611
- [Result] Zahiri M, Chen KM, Zhou H, Nguyen H, Workeneh BT, Yellapragada SV, Sada YH, Schwenk M, Najafi B. Using wearables to screen motor performance deterioration because of cancer and chemotherapy-induced peripheral neuropathy (CIPN) in adults - Toward an early diagnosis of CIPN. J Geriatr Oncol. 2019 Nov;10(6):960-967. doi: 10.1016/j.jgo.2019.01.010. Epub 2019 Jan 18. PMID 30665876
- See also: obstacle crossing exergame — https://www.youtube.com/watch?v=cYvNI7yfTiA